CLINICAL TRIAL: NCT02744170
Title: Effects of Supplemental Oxygen Delivery Via Demand Versus Continuous Flow in Hypoxemic COPD Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Schön Klinik Berchtesgadener Land (Other)
Responsible Party: Principal Investigator, Klaus Kenn, Prof. Dr. Klaus Kenn, Schön Klinik Berchtesgadener Land
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: O2-Demand-Study
Record Dates: First submitted 2016-03-08; First posted 2016-04-20 (Estimated); Last update posted 2019-01-22 (Actual); Status verified 2019-01

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; Incremental Shuttle Walk Test; Endurance Shuttle Walk Test; oxygen therapy
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- COPD patients with delivery order 1, 2, 3 (Experimental): Patients on long-term oxygen therapy will perform 3 Endurance Shuttle Walk Tests on three consecutive days with one of three different Oxygen delivery devices.
  Interventions: Device: 1 continuous flow oxygen supplementation; Device: 2 demand delivery liquid oxygen supplementation; Device: 3 demand delivery oxygen supplementation via concentrator
- COPD patients with delivery order 2,3, 1 (Experimental): Patients on long-term oxygen therapy will perform 3 Endurance Shuttle Walk Tests on three consecutive days with one of three different Oxygen delivery devices.
  Interventions: Device: 1 continuous flow oxygen supplementation; Device: 2 demand delivery liquid oxygen supplementation; Device: 3 demand delivery oxygen supplementation via concentrator
- COPD patients with delivery order 3, 2, 1 (Experimental): Patients on long-term oxygen therapy will perform 3 Endurance Shuttle Walk Tests on three consecutive days with one of three different Oxygen delivery devices.
  Interventions: Device: 1 continuous flow oxygen supplementation; Device: 2 demand delivery liquid oxygen supplementation; Device: 3 demand delivery oxygen supplementation via concentrator
- COPD patients with delivery order 1, 3, 2 (Experimental): Patients on long-term oxygen therapy will perform 3 Endurance Shuttle Walk Tests on three consecutive days with one of three different Oxygen delivery devices.
  Interventions: Device: 1 continuous flow oxygen supplementation; Device: 2 demand delivery liquid oxygen supplementation; Device: 3 demand delivery oxygen supplementation via concentrator
- COPD patients with delivery order 2, 1, 3 (Experimental): Patients on long-term oxygen therapy will perform 3 Endurance Shuttle Walk Tests on three consecutive days with one of three different Oxygen delivery devices.
  Interventions: Device: 1 continuous flow oxygen supplementation; Device: 2 demand delivery liquid oxygen supplementation; Device: 3 demand delivery oxygen supplementation via concentrator
- COPD patients with delivery order 3, 1, 2 (Experimental): Patients on long-term oxygen therapy will perform 3 Endurance Shuttle Walk Tests on three consecutive days with one of three different Oxygen delivery devices.
  Interventions: Device: 1 continuous flow oxygen supplementation; Device: 2 demand delivery liquid oxygen supplementation; Device: 3 demand delivery oxygen supplementation via concentrator

INTERVENTIONS:
Device: 1 continuous flow oxygen supplementation — This oxygen Supplementation is used in special order
  Other Names: Companion 1000 Chart Industries, Inc. Garfield Heights, USA
Device: 2 demand delivery liquid oxygen supplementation — This oxygen Supplementation is used in special order
  Other Names: Caire Spirit 300 Chart Industries, Inc. Garfield Heights
Device: 3 demand delivery oxygen supplementation via concentrator — This oxygen Supplementation is used in special order
  Other Names: one oxygen concentrator, Inogen, Goleta, CA, USA

SUMMARY:
Oxygen supplementation has been proven to be effective in hypoxemic COPD patients by increasing oxygenation and reducing dyspnea. In clinical practice there are three common oxygen delivery systems used: continuous oxygen flow (CF), demand oxygen delivery with liquid oxygen (DDL) and demand oxgen delivery with portable oxygen concentrator (DDC). The CF involves considerable wastage of oxygen because oxygen is supplied during in- and exhalation. Demand oxygen delivery saves oxygen and results in a comparable oxygen saturation at rest in COPD patients. However, it is unknown, if oxygen supplementation via demand oxygen delivery is also sufficient during exercise in hypoxemic COPD patients. In addition, it has to be considered that the lower weight of demand oxygen delivery system might enable patients for higher physical activity level and mobility in daily life.

The effects of These three oxygen delivery systems shall be investigated by a randomized, controlled cross-over Trial. Every patient has to perform an Incremental Shuttle Walk Test and three Endurance Shuttle Walk Tests with three different oxygen supplementation (via CF, DDL or DDK) in randomized order.

DETAILED DESCRIPTION:
The Principal Investigator will inform each patient about procedure, content and measurements of the study. It is obligatory that each patient participating in the study gives a written informed consent.

Following an initial incremental shuttle walk test (ISWT) in order to determine the individual maximum capacity, patients will perform three endurance shuttle walk tests (ESWT) at 85% of the maximal pace. In randomized order, patients will complete one ESWT on CF, one on DDL (liquid oxygen) and one on DDC (portable oxygen concentrator). The time between the three ESWTs will be 24 hours in order to give enough time for regeneration. All patients will use the same oxygen devices (CF: Companion 1000 (CE 0050), Chart Industries, Inc. Garfield Heights, Ohio, USA; DD [liquid oxygen]: Caire Spirit 300 (CE 0029), Chart Industries, Inc. Garfield Heights, Ohio, USA), DD [portable concentrator]: Inogen G2, California, USA) and will carry the oxygen device in a backpack. Continuous oxygen flow in liter per minute will be compared to the level of demand delivery (e.g.: 2 l/min CF will be compared to DD level 2).

ELIGIBILITY:
Inclusion Criteria:

* COPD patients (GOLD stage III to IV) with hypoxemia at rest or during exercise (paO2<60mmHg)
* Participation in an inpatient pulmonary rehabilitation program (Schön Klinik BGL)
* Written informed consent

Exclusion Criteria:

* General exclusion criteria for exercise tests, e.g. acute coronary syndrome, acute myo- or pericarditis, acute lung embolism, pulmonary infarction, acute uncontrolled heart insufficiency
* Signs of acute exacerbation
* Any orthopedic or neurological disabilities that prevent patient from walking

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Oxygen saturation at isotime of the endurance shuttle walk test (ESWT), compared between CF (liquid oxygen) and DD (liquid oxygen) | at baseline, at isotime of ESWT and at the end (maximal 20 min) of ESWT
  continuous transcutaneous recording during ESWT by Sentec-Digital-Monitor

SECONDARY OUTCOMES:
Breathing frequency | at baseline, at isotime of ESWT and at the end (maximal 20 min) of ESWT
  measured by Visionox
Inspiratory capacity | at baseline, at isotime of ESWT and at the end (maximal 20 min) of ESWT
  measured by Spiropalm
Heart rate | at baseline, at isotime of ESWT and at the end (maximal 20 min) of ESWT
  continuous transcutaneous recording during ESWT by Sentec-Digital-Monitor
Walking distance during ESWT | at baseline, at isotime of ESWT and at the end (maximal 20 min) of ESWT
  total distance walked during ESWT
dyspnea | at baseline, at isotime of ESWT and at the end (maximal 20 min) of ESWT
  assessed by modified Borg scale (0 to 10)
partial pressure of carbon dioxide | at baseline, at isotime of ESWT and at the end (maximal 20 min) of ESWT
  continuous transcutaneous recording during ESWT by Sentec-Digital-Monitor

CONTACTS AND LOCATIONS:
Overall Officials: Klaus Kenn, Prof. Dr., Principal Investigator — Philipps University Marburg
Locations (1):
- Klinikum Berchtesgadener Land, Schönau, Berchtesgardener Land, Germany

IPD SHARING:
Plan to Share IPD: No